CLINICAL TRIAL: NCT02784951
Title: Use of Blood and Plasma in Prehospital Haemorrhagic Shock - a Prospective, Observational Trial of Advanced Deployment of Blood Products in Norwegian Physician-staffed Helicopter Emergency Medical System
Brief Title: Use of Blood and Plasma in Norwegian Physician-staffed Helicopter Emergency Medical System
Acronym: ProHEMS
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Sykehuset Innlandet HF (Other); Oslo University Hospital (Other); Sorlandet Hospital HF (Other Government); St. Olavs Hospital (Other); Helse Forde (Other); Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/304/REK vest
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Hemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Erythrocyte Count; formycin diphosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single group: Patients in haemorrhagic shock needing volume replacement and receiving prehospital transfusion of blood products, either red blood cells (RBC), freeze dried plasma (FDP) or whole blood (WB).
  Interventions: Drug: Red blood cells (0Rh D-neg); Drug: Whole blood (O Rh D-neg K-neg); Drug: Freeze dried plasma (LyoPlas)

INTERVENTIONS:
Drug: Red blood cells (0Rh D-neg) — Fresh produced RBC
  Other Names: RBC
Drug: Whole blood (O Rh D-neg K-neg) — Fresh produced WB
  Other Names: WB
Drug: Freeze dried plasma (LyoPlas) — (LyoPlas N-w (German Red Cross)
  Other Names: FDP

SUMMARY:
The main objective of this study is to evaluate the use of RBC, FDP, WB in the treatment of exsanguinating patients by physician-staffed emergency medical services in Norway, with focus on prehospital transfusion complications and safety.

DETAILED DESCRIPTION:
This study evaluates prehospital transfusion therapy in exsanguinating patients treated by physician-staffed emergency medical services in Norway, with the following main questions:

I. Are out-of-hospital transfusions associated with an increase in adverse transfusion events compared to inhospital transfusions?

II. Is out-of-hospital physician administration of plasma or blood products in exsanguinating patients feasible?

III. Are patients in need of blood product transfusion possible to identify and transfuse in the prehospital phase/environment?

IV. Are out-of-hospital transfusion practices associated with increased waste of blood products?

All patients in haemorrhagic shock needing volume replacement and receiving prehospital transfusion of blood products will be included, if they fulfill the listed criteria below:

* Patients with mechanism of injury compatible with severe haemorrhage and/or haemorrhagic shock (e.g. penetrating torso injury, visible massive bleeding)
* Radial pulse > 100 beats/min or absent/weak radial pulse
* Systolic blood pressure (SBP) < 90 mmHg
* Altered mental status (reduced GCS) in the absence of head injury or known intoxication

Patients with known previous serious allergic reactions to blood product transfusions or patients who refuse blood products on religious grounds (e.g. Jehovah´s Witness) will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* All patients in haemorrhagic shock needing volume replacement and receiving prehospital transfusion of blood products according to listed indicators below:

  * Patients with mechanism of injury compatible with severe haemorrhage and/or haemorrhagic shock (e.g. penetrating torso injury, visible massive bleeding)
  * Radial pulse > 100 beats/min or absent/weak radial pulse
  * Systolic blood pressure (SBP) < 90 mmHg
  * Altered mental status (reduced GCS) in the absence of head injury or known intoxication

Exclusion Criteria:

* Patients with known previous serious allergic reactions to blood product transfusions
* Patients who refuse blood products on religious grounds, e.g. Jehovah´s Witness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (pediatric and adult) in haemorrhagic shock needing volume replacement and receiving prehospital transfusion of blood products by treating physician staffed emergency medical services.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
adverse transfusion reactions | 24 hours
  Fraction of patients with suspected adverse transfusion reactions after administration of plasma and/or blood products.
patients included | 24 hours
  Fraction of patients fulfilling inclusion criteria with prehospital administration of blood products
units not used | 24 hours
  Fraction of prepared plasma or blood units not used.

SECONDARY OUTCOMES:
Number of adverse events | 24 hours
  Number of adverse events (e.g. transfusion related complications or reactions (first 24 hrs))
Type of adverse events | 24 hours
  Type of adverse events (e.g. transfusion related complications or reactions (first 24 hrs))
number of transfusion | 24 hours
  Number of transfusions given prehospital and inhospital (first 24 hrs)
type of transfusion | 24 hours
  type of transfusions given prehospital and inhospital (first 24 hrs)
Systolic blood pressure (SBP) | 24 hours
  Systolic blood pressure (SBP) on scene and at admission hospital
heart rate (HR) | 24 hours
  heart rate (HR) on scene and at admission hospital
Glasgow Coma Score (GCS) | 24 hours
  Glasgow Coma Score (GCS) on scene and at admission hospital
Respiratory rate (RR) | 24 hours
  Respiratory rate (RR) on scene and at admission hospital
Pulse oximeter (SPO2) | 24 hours
  Pulse oximeter (SPO2) on scene and at admission hospital
response time (minutes) | 24 hours
  Physician staffed emergency medical services response (in minutes) from dispatch to arrival on-scene
on-scene time (minutes) | 24 hours
  Time (in minutes) from emergency medical services arrival on-scene until patients leaves the scene or is pronounced dead on-scene
transport time (minutes) | 24 hours
  Time (in minutes) from the patients leaves the scene until patient arrives in hospital
Number of surgical interventions | 24 hours
  Number of surgical interventions (first 24 hrs)
Type of surgical interventions | 24 hours
  type of surgical interventions (first 24 hrs)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Klausen, MD, Study Director — Medical Director, Kirurgisk Serviceklinikk, Haukeland Universitetssykehus
Locations (9):
- Norway (9):
  - Sørlandet Hospital HF, Arendal
  - Haukeland University Hospital, Bergen
  - Innlandet Hospital Trust, Brumunddal
  - Vestre Viken Hospital Trust, Drammen
  - Helse Førde, Førde
  - Oslo University Hospital, Oslo
  - Helse Stavanger HF, Stavanger
  - University Hospital of North Norway, Tromsø
  - St Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sunde GA, Bjerkvig C, Bekkevold M, Kristoffersen EK, Strandenes G, Bruserud O, Apelseth TO, Heltne JK. Implementation of a low-titre whole blood transfusion program in a civilian helicopter emergency medical service. Scand J Trauma Resusc Emerg Med. 2022 Dec 9;30(1):65. doi: 10.1186/s13049-022-01051-z. PMID 36494743